CLINICAL TRIAL: NCT02933476
Title: Vibrotactile Stimulation in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: John A Blume Foundation (Unknown)
Responsible Party: Principal Investigator, Helen M. Bronte-Stewart, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 35238
Record Dates: First submitted 2016-07-08; First posted 2016-10-14 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vibrotactile Stimulation Treatment (Experimental): All patients will receive the vibrotactile stimulation treatment. No deception will be used.
  Interventions: Device: Vibrotactile Stimulation

INTERVENTIONS:
Device: Vibrotactile Stimulation — The tactile stimulator is being tested for an off-label use as treatment for Parkinson's disease. There are nodes embedded into the fingertips of gloves that gently vibrate in an alternating pattern. The sensation is similar to the feeling of a phone vibrating. This is a non-significant risk device.

SUMMARY:
The purpose of this study is to examine the possibility of a new, non-invasive, non-drug treatment for Parkinson's disease. The treatment involves gentle vibratory stimulation delivered to the fingertips (called 'vibrotactile stimulation'). Along with the treatment, participants will also undergo kinematic testing.

DETAILED DESCRIPTION:
Patient will be phone screened and/or have a physical and neurological examination to determine if it is appropriate for them to participate in this study. This testing includes the Unified Parkinson's Disease Rating Scale, Part III (UPDRS III). Research assistants will explain the study and obtain informed consent. There will be three consecutive days of testing, as well as 2 follow up visits at 1 and 4 weeks. Visits include the following: Patients will have sensors put on their hands, feet, and chest. These sensors measure their movement while they perform kinematic tasks such as forward walking, wrist movements, and the UPDRS III. Patients will also be given vibrotactile stimulation for a total of 4 hours throughout the day. During this time, patients will be provided with books/movies as entertainment, and they may move around freely. Patients will also be asked to complete several questionnaires throughout the visits about their Parkinson's symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years of age.
2. Speaks and understands English.
3. A diagnosis of idiopathic Parkinson's disease, Hoehn and Yahr Stage II or III
4. Able and willing to come to study visits (3 consecutive days, as well as 2 follow up visits, at 1 and 4 weeks)
5. Able and willing to stop therapy during the daytime for the days they come to the clinic for the study.
6. Have improvement in motor signs ON versus OFF dopaminergic medication.
7. If on medication, the patient should be on stable doses of Sinemet and/or Stalevo (Carbidopa/Levodopa Parkinson's medication) as part of their medicinal regimen (Patient does not need to be on medication to be included in the study).

Exclusion Criteria:

1. Subjects, who are pregnant, are capable of becoming pregnant, or who are breast feeding.
2. Subjects with very advanced Parkinson's disease, Hoehn and Yahr stage IV on medication (non-ambulatory).
3. Have significant cognitive impairment and/or dementia, as determined by a neurologist at the Stanford Movement Disorders Clinic.
4. Have an implanted electronic device such as a cardiac pacemaker/defibrillator or medication pump.
5. Subjects who have an inability to comply with study follow-up visits.
6. Subjects who are unable to understand or sign the informed consent.
7. Have an MRI showing focal brain lesions that could indicate a non-idiopathic movement disorder.
8. Have an active infection.
9. Require diathermy, electroconvulsive therapy (ECT), or transcranial magnetic stimulation (TMS) to treat a chronic condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Bronte-Stewart, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford Movement Disorders Clinic, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adamchic I, Hauptmann C, Barnikol UB, Pawelczyk N, Popovych O, Barnikol TT, Silchenko A, Volkmann J, Deuschl G, Meissner WG, Maarouf M, Sturm V, Freund HJ, Tass PA. Coordinated reset neuromodulation for Parkinson's disease: proof-of-concept study. Mov Disord. 2014 Nov;29(13):1679-84. doi: 10.1002/mds.25923. Epub 2014 Jun 28. PMID 24976001
- [Background] Tass PA. A model of desynchronizing deep brain stimulation with a demand-controlled coordinated reset of neural subpopulations. Biol Cybern. 2003 Aug;89(2):81-8. doi: 10.1007/s00422-003-0425-7. Epub 2003 Jul 14. PMID 12905037

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 6 subjects were enrolled, but data only collected for 5 subjects. (1 subject was enrolled but no baseline data was collected due to illness)
Period: Overall Study
Arm/Group | Vibrotactile Stimulation Treatment
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vibrotactile Stimulation Treatment
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 5
Unified Parkinson's disease Rating Scale, Part III [Mean (Standard Deviation); unit: units on a scale] — The Unified Parkinson's disease Rating Scale (UPDRS) has a total of four parts. We have used Part III which is the motor examination portion, excluding rigidity and speech. The total score ranges from 0 to 108. 108 represents the worst disability and 0 no disability
  units on a scale | 21 (12.8)
Disease Duration [Mean (Standard Deviation); unit: years] | 5.718 (2.694)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reporting Any Adverse Effects
Description: Questionnaire asks patients to record any adverse effects they experienced.
Time Frame: 1 Month
Measure: Count of Participants; unit: Participants
Arm/Group | Vibrotactile Stimulation Treatment
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Unified Parkinson's Disease Rating Scale, Part III
Description: We used the motor portion of the Unified Parkinson's disease Rating Scale (UPDRS) and excluded rigidity and speech from the assessment. Overall range of the score for the motor portion (excluding rigidity and speech) range from 0 to 108, where 0= best possible outcome and 108= worst possible outcome.
Time Frame: 1 Month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vibrotactile Stimulation Treatment
Number analyzed (Participants) | 5
units on a scale
  UPDRS III at Baseline | 21 (12.8)
  UPDRS III at 1 week from baseline | 21.8 (11.7)
  UPDRS III at 4 weeks from baseline | 20.8 (14.8)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation Treatment; We compared off therapy UPDRS III scores at baseline to one and four weeks after stimulation; Test type: Superiority; p > 0.05, ANOVA

3. Secondary Outcome: Root Mean Square Velocity
Description: Using gyroscopes to track patient movement testing, root mean square velocity (Vrms) of of the wrist during repetitive wrist flexion extension task was obtained.
Time Frame: 1 Month
Population: One out of the five patients was on medication so was excluded from analysis.
Measure: Mean (Standard Deviation); unit: deg/s
Arm/Group | Vibrotactile Stimulation Treatment
Number analyzed (Participants) | 4
deg/s
  Average Vrms at baseline | 350.637 (140.222)
  Average Vrms at 1 month | 456.736 (156.634)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation Treatment; Test type: Superiority; p = 0.008, ANOVA

4. Secondary Outcome: Gait Asymmetry
Description: Using data collected from inertial measurement unit (IMU) sensors on subject, we were able to measure gait asymmetry. For each subject, the swing time (SW) was calculated and averaged across strides for the left and right legs (SWL and SWR). We obtained gait asymmetry using the following: 100 x /ln(SWR/SWL)/. 0 marks perfect symmetry and greater values higher asymmetry. There is no maximum limit.
Time Frame: 1 Month
Population: One out of the five patients was on medication so was excluded from analysis.
Measure: Mean (Standard Deviation); unit: arb.units
Arm/Group | Vibrotactile Stimulation Treatment
Number analyzed (Participants) | 4
arb.units
  Average gait asymmetry at 1 month | 4.53 (5.51)
  Average gait asymmetry at baseline | 8.51 (5.66)
Statistical Analysis 1: Comparison: Vibrotactile Stimulation Treatment; Test type: Superiority; p < 0.001, ANOVA

ADVERSE EVENTS:
Time Frame: 1 month
Description: Adverse Events Questionnaire was given to participants following each visit
Arm/Group | Vibrotactile Stimulation Treatment
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No